CLINICAL TRIAL: NCT00319826
Title: Virulence Determinants in Staphylococcus Aureus Bacteremia
Brief Title: Virulence Determinants in S Aureus Bacteremia
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00014073; 04-087
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Bacteremia
Keywords: Staphylococcus aureus, S. aureus, bacteremia, sepsis
MeSH Terms: conditions — Bacteremia; Staphylococcal Infections; Sepsis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Subjects with Staphylococcus Bacteremia
- 2: Healthy (Non-infected) Control Subjects in the Nasal Carriage Group
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study with no intervention
  Other Names: Observational Study
  Groups: 2

SUMMARY:
The purpose of this study is to investigate why some people develop life-threatening infections caused by the bacteria Staphylococcus aureus, while other people do not. It is possible that the infectious ability of the bacteria can determine whether an infection develops and its severity. The investigators will look at old blood and nasal specimens collected from 1000 adults who had S. aureus infections and who were hospitalized at Duke University Medical Center. Previously collected health information regarding these patients and the specific bacterial traits in the samples will be studied. Eventually this information may be used to help treat and prevent S. aureus infection.

DETAILED DESCRIPTION:
The purpose of this study is to more thoroughly investigate the impact of bacterial genetic characteristics on the outcome of patients with S. aureus bacteremia (SAB). The investigators will address salient aspects of bacterial virulence using strong collaborative relationships with authorities in bacterial genetics and genomics. The overall hypothesis of this investigation is that distinct bacterial virulence determinants influence the severity of S. aureus infection. The specific hypothesis is that virulence determinants associated with clinical outcome of S. aureus infection segregate into clonal groups, identified by Multilocus Sequence Typing (MLST), and can be localized in the genome by comparative genetic hybridization (CGH). The investigators have established the following aims to pursue this hypothesis. Specific Aim 1: Define the allelic diversity of S. aureus bloodstream isolates using MSLT. Allelic profiles among the 1000 isolates will be compared using the program BURST (Based Upon Related Sequence Type), and relatedness of lineages in the overall collection will be defined. Specific Aim 2: Define the genomic diversity of S. aureus bloodstream isolates using CGH. Using MLST results, a subset of 200 isolates will be selected to undergo further study. These ~200 isolates will form a unique collection hereafter referred to as the SAGA (S. aureus genomic analysis) collection. The genomic diversity of the SAGA subset will be defined using CGH. Specific Aim 3: Correlate MLST and CGH results, MLST and clinical outcome, and CGH, and clinical outcome, and make SAGA isolates available to the scientific community. In this Specific Aim, the discriminate ability of MLST and CGH will be compared among the SAGA subset isolates undergoing both assays. The association between bacterial clonality and clinical outcome will be considered among 1000 S. aureus isolates collected from adults at Duke University Medical Center who had S. aureus infections undergoing MLST. The association between clinical outcome and the presence or absence of virulence factors and pathogenicity islands in the S. aureus genome will also be considered among the 200 SAGA subset isolates undergoing CGH. The products of this study will include an increased understanding of genetic diversity in S. aureus and the role of this genetic diversity on determining the severity of infections caused by S. aureus. The full value of the current proposal also includes the potential future benefit to the research community as a whole if associations between pathogen genotype and clinical outcome, only possible to identify using such a large and clinically well-characterized collection of isolates, can be defined. To amplify these potential downstream dividends, the final goal of Specific Aim 3 will be to make SAGA subset isolates, corresponding MLST types, and CGH profiles available to the scientific community through the repository maintained by the Network for Antimicrobial Resistance in S. aureus (NARSA). The long-term objectives of this project are to: (1) identify bacterial genes contributing to the severity of infection in isolates from a large cohort of patients with SAB; and (2) ultimately use these genes to identify novel interventions for the control of S. aureus pathogenesis by investigating genes that govern the virulence of this emerging pathogen. Culture-confirmed SAB nasal carriage isolates and/or bloodstream bacterial isolates previously collected from 1000 inpatient adults at Duke University Medical Center will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (>= 18 years) with culture-confirmed Staphylococcus aureus bacteremia (SAB). Patients with SAB transferred to Duke University Medical Center are eligible if speculation and antibiotic susceptibilities are confirmed by the Duke Clinical Microbiology Laboratory.
2. Absolute neutrophil count of > 1000 cells/cubic millimeter at the time that the initial positive blood culture is obtained.
3. Patient or patient's representative provides signed informed consent allowing study participation.

Exclusion Criteria:

1. Prior enrollment of patient in this investigation (to ensure statistical independence of observations).
2. Staphylococcus aureus bacteremia (SAB) that is not confirmed by culture and speciation at the Duke Clinical Microbiology Laboratory.
3. Outpatient status.
4. Isolation of any pathogen other than S. aureus from bloodstream.
5. Inability of patient or patient's representative to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bacterial strains are used from patients with particular syndromes (e.g. nasal carraige, endocarditis, osteomylitis) that were be identified using the Bloodstream Infections Registry. No new subjects was or will be enrolled within the current investigation.
Sampling Method: Non-Probability Sample
Enrollment: 1354 (Actual)
Dates: Start 2004-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Cure vs. recurrence of Staph infection vs. death | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vance G. Fowler, MD, Principal Investigator — Duke UMC
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States